CLINICAL TRIAL: NCT04592705
Title: Measurement of IL-6 and Secondary Inflammatory Markers Before and After Therapeutic Plasma Exchange (TPE) in Hospitalized Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Larkin Community Hospital (Other)
Responsible Party: Principal Investigator, Michael Talalaev, M.D., D.O., Principal Investigator, Larkin Community Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: LCH-1-092020
Record Dates: First submitted 2020-10-07; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: COVID-19
Keywords: therapeutic plasma exchange; covid19; coronavirus
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Plasma Exchange

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Therapeutic plasma exchange (Experimental)
  Interventions: Device: Therapeutic plasma exchange

INTERVENTIONS:
Device: Therapeutic plasma exchange — TPE is the process of plasmapheresis, an invasive procedure separating plasma from red blood cells using centrifuge-based devices.
  Filtration involves the insertion of a central venous catheter in the internal jugular, femoral or subclavian vein after which blood is drawn from the patient's circulation and transferred to a filter that separates the plasma from blood cells. Thereafter, the plasma extracted is substituted with human albumin and/or FFP.

SUMMARY:
Given the current lack of an effective drug or therapy, a clinical trial to better understand the safety and efficacy of therapeutic plasma exchange (TPE) in COVID-19 patients is urgently needed. The goal of this trial is to study the efficacy and safety of TPE therapy in subjects with moderate to severe COVID-19 by determining the morbidity and mortality after TPE therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with moderate-severe COVID-19 infection including early acute lung injury (ALI)/early acute respiratory distress syndrome (ARDS)
2. Able to provide Informed Consent signed by the subject or by the subject's legal or healthcare proxy.
3. Admitted to the participating facilities as listed above (Larkin South Miami Hospital, Larkin Palm Springs Hospital).
4. Subjects between 18 and 69 years of age.
5. If female, subjects that have a negative result in a quantitative b-HCG blood test if they are within reproductive age.
6. A positive COVID-19 test via nasopharyngeal swab RT-PCR.
7. Agree to not participate in another clinical trial during the study period.

Exclusion Criteria:

1. Under 18 years of age or older than 69 years of age.
2. Severe disease, defined as:

   i. dyspnea ii. respiratory frequency ≥ 30/min iii. blood oxygen saturation ≤ 93% iv. partial pressure of arterial oxygen to fraction of inspired oxygen ratio < 300, and/or v. lung infiltrates > 50% within 24 to 48 hours;
3. Life-threatening disease, defined as:

   i. respiratory failure ii. septic shock, and/or iii. multiple organ dysfunction or failure
4. Unable to provide informed consent or decline to consent.
5. Sequential Organ Failure Assessment (SOFA) score of 12 or above.
6. Hemodynamic instability, sepsis, or other conditions causing inability to tolerate fluid shifts
7. Inability to tolerate central line placement
8. Allergy to FFP or albumin
9. Severe hypocalcemia
10. Patients with heparin allergies should not receive heparin as an anticoagulant during plasmapheresis
11. Patients taking angiotensin-converting enzyme (ACE) inhibitors are advised to stop taking the medication for at least 24 hours before starting plasmapheresis
12. Active or recent bleeding (unless controlled for >48 hours).
13. Thrombocytopenia (≤25,000/L).
14. Advanced cirrhosis with a history of esophageal varices.
15. Chronic kidney disease requiring hemodialysis.
16. Active solid or non-solid malignancy or Lymphoma within the last 2 years.
17. Heart failure (NYHA class III or IV).
18. HIV infection (AIDS criteria), a history of immunodeficiency, or subject is currently receiving immunosuppressive therapy.
19. Women of childbearing age who are pregnant or intend to become pregnant during the study period.
20. Known history of chromosomal or genetic abnormalities.
21. History of hypersensitivity or any kind of adverse reaction to blood products.
22. Contraindication to transfusion of blood products, or refusal due to religious/personal reasons.
23. Any kind of drug or alcohol dependence that would interfere with adherence to the study requirements.
24. Already part of this trial, recruited at a different hospital.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-09-11 (Actual); Primary Completion 2021-08-30 (Estimated); Study Completion 2021-08-30 (Estimated)

PRIMARY OUTCOMES:
Time to clinical status downgrade or discharge. | 60 days
  Clinical improvement will be defined as a point reduction in subjects' clinical status on the 8-point WHO ordinal scale for clinical improvement or discharge from the hospital, whichever comes first.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Talalaev, D.O., Principal Investigator — Larkin Community Hospital
Locations (1):
- Larkin Community Hospital, South Miami, Florida, United States

DOCUMENTS (1):
  • Informed Consent Form (2020-10-07): https://cdn.clinicaltrials.gov/large-docs/05/NCT04592705/ICF_000.pdf